CLINICAL TRIAL: NCT03889626
Title: A Phase III Study of Comparing the Maintenance Treatment of Apatinib, Capecitabine and Observation After First-line Therapy in Advanced Gastric Cancer
Brief Title: The Maintenance Treatment of Apatinib/Capecitabine Versus Observation in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, Principal Investigator and Clinical Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Apa/Cap maintenance in GC
Record Dates: First submitted 2019-03-17; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Stomach Neoplasms; Gastrointestinal Neoplasms; Stomach Diseases; Digestive System Neoplasms; Capecitabine; Apatinib; Neoplasms; Molecular Mechanisms of Pharmacological Action
Keywords: Capecitabine; Apatinib; Maintenance Treatment; Advance Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Neoplasms; Stomach Diseases; Digestive System Neoplasms; Neoplasms | interventions — apatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Apatinib (Experimental): In this arm, patients will receive a daily oral treatment with Apatinib 500mg.
  Interventions: Drug: Apatinib
- Capecitabine (Experimental): In this arm , patients will receive capecitabine 1000mg/m2 twice for 14 days, and repeat every 3 weeks.
  Interventions: Drug: Capecitabine
- Observation (No Intervention): In this arm, no additional treatment will be given, and patients will be followed up at regular time

INTERVENTIONS:
Drug: Apatinib — Apatinib: 500mg qd po, q4w
  Arms: Apatinib
Drug: Capecitabine — Capecitabine: 1000mg/m2 bid po, d1-14, q3w
  Arms: Capecitabine

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of the maintenance treatment of Apatinib/Capecitabine after fluorouracil and platinum based first-line chemotherapy in advanced gastric cancer.

DETAILED DESCRIPTION:
Up to now, whether maintenance therapy after first line treatment can bring survival benefits to patients with advanced gastric cancer is unknown, and let alone which drug is most suitable. Our study is designed to prove whether the maintenance treatment of Apatinib or Capecitabine are better than observation after fluorouracil/platinum based first-line chemotherapy in advanced gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic gastric or gastroesophageal junction adenocarcinoma
* ECOG PS 0-2
* At least one measurable or evaluable lesion in the first-line chemotherapy
* The fist line treatment should be 5-FU based regimen (e.g. ECF/EOF/EOX/FOLFOX/XELOX/XP) , and patients should received 6 cycles (3-week regimen) or 12 cycles (2-week regimen) treatment with the efficacy of non-PD
* The time from the last cycle treatment to the enrollment cannot exceed 6 weeks
* Adequate hepatic, renal, heart, and hematologic functions (platelets ≥75×109/L, neutrophil ≥1.5×109/L, hemoglobin ≥80 g/L, serum creatinine ≤1.5mg/dl, total bilirubin ≤1.5mg/dl, and serum transaminase ≤2.5× the ULN)

Exclusion Criteria:

* Received 2 or more regimens for palliative chemotherapy
* Pregnant or lactating women
* Concurrent cancer, or history of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Uncontrolled brain, or leptomeningeal involvement, complete intestinal obstruction
* Clinically significant active bleeding, OB 2+ or higher
* Patients with locally advanced gastric cancer who are scheduled to receive radiotherapy
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months or high risk/uncontrolled arrhythmia
* Uncontrolled significant comorbid conditions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — no younger than 18 year-old
Enrollment: 242 (Estimated)
Dates: Start 2019-03-22 (Estimated); Primary Completion 2022-03-22 (Estimated); Study Completion 2024-03-22 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | six weeks
  PFS is calculated from the time of randmization to disease progression or death whichever happen first

SECONDARY OUTCOMES:
Overall Survival (OS) | six weeks
  OS is calculated from the time of randmization to death

OTHER OUTCOMES:
Quality of Life (QoL) | six weeks
  we will use EORTC QLQ-C30 to evaluate QoL.
Adverse Events | six weeks
  we will use CTC AE4.0 to evaluate adverse events.

IPD SHARING:
Plan to Share IPD: No